CLINICAL TRIAL: NCT06240819
Title: Comparison of Cross Body and Sleeper Stretch on Pain, Range of Motion and Functional Performance in Cricket Bowlers With Glenohumeral Internal Rotation Deficiency(GIRD).
Brief Title: Cross Body vs Sleeper Stretch on Pain, Range of Motion and Functional Performance in Cricket Bowlers.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0447
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Pain; Range of Motion; Physical Functional Performance
Keywords: Cross body Stretch; Sleeper stretch; Functional Performance; Glenohumeral internal rotation deficit; Cricket bowlers
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: randomized clinical trail
Who Masked: Outcomes Assessor
Masking Description: the assessor who will take the readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleeper Stretch (Other): Sleeper stretch in a side lying position in 90o abduction, elbow at 90o flexion and then performing shoulder IR for three sets with three repetitions.
  Interventions: Other: Sleeper Stretch
- Cross Body Stretch (Other): cross-body stretch will be done in sitting position. Three sets of the each stretch position would be held for 30 seconds with a 1 minute break between sets.
  Interventions: Other: Cross Body Stretch

INTERVENTIONS:
Other: Sleeper Stretch — They will receive three sessions a week for four weeks. In a session three sets with three repetitions of sleeper stretch in a side lying position
  Arms: Sleeper Stretch
Other: Cross Body Stretch — They will receive three sessions a week for four weeks. In a session, three sets with three repetitions of cross-body stretch will be done in sitting position.
  Arms: Cross Body Stretch

SUMMARY:
The study is randomized and single-blinded. Ethical approval is taken from ethical committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelope method by Non-probability Convenient random sampling technique. Subjects in Group A will receive sleeper stretch in a side lying position. Group B will receive cross-body stretch will be done in sitting position

DETAILED DESCRIPTION:
The objective of the study is to determine the comparison of sleeper stretch and cross body stretch on pain, range of motion and functional performance in cricket bowlers with GIRD. The study is randomized and single-blinded. Ethical approval is taken from ethical committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelope method by Non-probability Convenient random sampling technique. Subjects in Group A will receive sleeper stretch in a side lying position. Group B will receive cross-body stretch will be done in sitting position. A universal goniometer, Upper limb functional index (UEFI) scale and Numeric pain rating scale (NPRS) will be used at the baseline and after the completion of treatment at 6 weeks.

The data will be analyzed by SPSS, version 25. Statistical significance is P=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 30years,
* Both male and female,
* >10% IR deficit,
* >25% IR deficit related to contralateral limb,
* Athletes one year of regular practice,
* Lift off test for shoulder internal rotation positive.

Exclusion Criteria:

* Non players,
* Any nerve lesions of upper limb,
* Players with history of shoulder pain or fracture or dislocation in less than twelve months

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain | pre and 6 weeks post interventional
  Numeric pain rating scale (NPRS) will be used to assess pain.
Range of motion | pre and 6 weeks post interventional
  A universal goniometer will be used to measure ROM
Functional Performance | pre and 6 weeks post interventional
  upper extremity functional index (UEFI) scale to assess functional performance

CONTACTS AND LOCATIONS:
Overall Officials: Sitara Jabeen, DPT, Principal Investigator — Study Principal Investigator
Locations (1):
- Pakistan sports board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giles K, Musa I. A survey of glenohumeral joint rotational range and non-specific shoulder pain in elite cricketers. Phys Ther Sport. 2008 Aug;9(3):109-16. doi: 10.1016/j.ptsp.2008.03.002. Epub 2008 May 9. PMID 19083711
- [Background] Rose MB, Noonan T. Glenohumeral internal rotation deficit in throwing athletes: current perspectives. Open Access J Sports Med. 2018 Mar 19;9:69-78. doi: 10.2147/OAJSM.S138975. eCollection 2018. PMID 29593438
- [Background] Wilk KE, Hooks TR, Macrina LC. The modified sleeper stretch and modified cross-body stretch to increase shoulder internal rotation range of motion in the overhead throwing athlete. J Orthop Sports Phys Ther. 2013 Dec;43(12):891-4. doi: 10.2519/jospt.2013.4990. Epub 2013 Oct 30. PMID 24175603
- [Background] Aldridge R, Stephen Guffey J, Whitehead MT, Head P. The effects of a daily stretching protocol on passive glenohumeral internal rotation in overhead throwing collegiate athletes. Int J Sports Phys Ther. 2012 Aug;7(4):365-71. PMID 22893856
- [Background] Mine K, Nakayama T, Milanese S, Grimmer K. Effectiveness of Stretching on Posterior Shoulder Tightness and Glenohumeral Internal-Rotation Deficit: A Systematic Review of Randomized Controlled Trials. J Sport Rehabil. 2017 Jul;26(4):294-305. doi: 10.1123/jsr.2015-0172. Epub 2016 Aug 24. PMID 27632891
- [Background] Johnson JE, Fullmer JA, Nielsen CM, Johnson JK, Moorman CT 3rd. Glenohumeral Internal Rotation Deficit and Injuries: A Systematic Review and Meta-analysis. Orthop J Sports Med. 2018 May 22;6(5):2325967118773322. doi: 10.1177/2325967118773322. eCollection 2018 May. PMID 29845083
- [Background] Dutton M, Tam N, Divekar N, Prins D, Gray J. The association between gird and overhead throwing biomechanics in cricket. J Biomech. 2021 Sep 20;126:110658. doi: 10.1016/j.jbiomech.2021.110658. Epub 2021 Jul 29. PMID 34358903
- [Background] Moradi M, Hadadnezhad M, Letafatkar A, Khosrokiani Z, Baker JS. Efficacy of throwing exercise with TheraBand in male volleyball players with shoulder internal rotation deficit: a randomized controlled trial. BMC Musculoskelet Disord. 2020 Jun 13;21(1):376. doi: 10.1186/s12891-020-03414-y. PMID 32534582